CLINICAL TRIAL: NCT05037994
Title: Ultrasound Guided Continuous Suprascapular Nerve Block With Oral Gabapentin For Pain Management In Patients With Frozen Shoulder
Brief Title: Suprascapular Nerve Block With Oral Gabapentin For Pain Management In Frozen Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Amr Shaaban Elshafei, AMR SHAABAN ELSHAFEI, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 6909
Record Dates: First submitted 2021-09-03; First posted 2021-09-08 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Pain, Shoulder
MeSH Terms: conditions — Shoulder Pain | interventions — Bupivacaine; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (C Group) (Placebo Comparator): Patients will receive continuous US suprascapular nerve block only.
  Interventions: Procedure: Ultrasound Guided Continuous Suprascapular Nerve Block With methyl prednisolone and marcaine
- Gabapentin Group (G Group) (Experimental): Patients will receive continuous US suprascapular nerve block with oral gabapentin 300 mg once daily at bed time.
  Interventions: Procedure: Ultrasound Guided Continuous Suprascapular Nerve Block With methyl prednisolone and marcaine

INTERVENTIONS:
Procedure: Ultrasound Guided Continuous Suprascapular Nerve Block With methyl prednisolone and marcaine — The high frequency linear ultrasound transducer (Sonosite 6-13 MHz) in a transverse orientation will be placed over the scapular Spine.
  Moving the transducer cephalad the suprascapular fossa will be identified. 18 gauge touhy needle will be inserted in plane after subcutaneous local anesthesia infiltration with 1 ml lidocaine 2% Real-time imaging will be used to direct injection of 2 ml lidocaine 2% to test perineural spread of injectate after confirmation of the position of tip of needle injection of 40mg methyl prednisolone diluted in 5 ml bupivacaine 0.5% will be done through the needle to anesthetize the nerve and create space for catheter insertion. After catheter insertion another 2 ml lidocaine 2% will be injected through the catheter to confirm position perineural in the scapular notch. Lastly Catheter will be fixed via skin tunnel and secured with skin sutures and adhesive tap.
  Other Names: Oral gabapentin 300 mg at bed time in GG

SUMMARY:
The patients will be randomly allocated into two equal groups (each 20 patients) using sealed opaque numbered envelopes:

Control Group (C Group) : Patients receive continuous US suprascapular nerve block only.

Gabapentin Group (G Group) : Patients receive continuous US suprascapular nerve block with oral gabapentin 300 mg once daily at bed time.

Both groups compared as regard:

Visual Analogue Scale Range of passive and active movements Patients satisfaction complication related to block The total dose of diclofenac sodium

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≥ 18 Kg/m2 ≤ 30Kg/m2
* ASA I, II or III.
* Cooperative patients.

Exclusion Criteria:

* local infection at site of injection.
* coagulopathy
* previous history of mental disorders or chronic drug abuse (opioids, tranquilizers)
* known hypersensitivity to any of the drugs used in the study.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | 6 weeks
  10cm line where zero means no pain and ten means worse imaginary pain

SECONDARY OUTCOMES:
Range of passive and active movements | 6 weeks
  by goniometer
Patients satisfaction | 6 weeks
  by questionnaire with 3 degrees
  1. Fair
  2. Good
  3. Excellent

OTHER OUTCOMES:
The total dose of diclofenac sodium | 6 weeks
  Indicator for analgesia required

CONTACTS AND LOCATIONS:
Overall Officials: AHMAD S HEGAB, MD, Study Director — Assistant professor of Anesthesia & Surgical Intensive Care Faculty of Medicine - Zagazig University
Locations (1):
- Amr Shaaban Elshafei, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No